CLINICAL TRIAL: NCT04299516
Title: Safety of Single-stage, Two-team, Simultaneous Bilateral Total Knee Arthroplasty Compared to One-team: A Randomized Controlled Trial
Brief Title: Bilateral Simultaneous Total Knee Arthroplasty for Bilateral Gonarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Gökçer Uzer, Associate Professor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08.11.2017-71306642-050.01.04
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Bilateral Total Knee Arthroplasty; Gonarthrosis; Primary, Bilateral
Keywords: total knee arthroplasty; complication; safety; operative time
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-team SBA (Experimental): Two-team simultaneous bilateral total knee arthroplasty
  Interventions: Procedure: Two-team simultaneous bilateral total knee arthroplasty
- Single-team SBA (Active Comparator): Single-team simultaneous bilateral total knee arthroplasty
  Interventions: Procedure: Single-team simultaneous bilateral total knee arthroplasty

INTERVENTIONS:
Procedure: Two-team simultaneous bilateral total knee arthroplasty — Bilateral total knee arthroplasty can be performed in three different ways: single-stage, two-team simultaneous bilateral total knee arthroplasty; single-stage, one-surgeon, and two-stage bilateral total knee arthroplasty. Two surgeons will operate simultaneously on one side for two-team SBA.
  Arms: Two-team SBA
Procedure: Single-team simultaneous bilateral total knee arthroplasty — One surgeon will operate sequentially on both sides for one-surgeon SBA
  Arms: Single-team SBA

SUMMARY:
The effects of two-team and single-team simultaneous bilateral total knee arthroplasty (SBA) on peri- and postoperative complications are not clear. The investigators hypothesized that two-team SBA has lower early postoperative complication rates than single-surgeon SBA. Therefore, this prospective study compared minor and major complications for 90 days postoperatively between two-surgeon and single-surgeon SBA.

DETAILED DESCRIPTION:
Study Design:

This prospective randomized study was approved by our institution's Clinical Research Ethics Committee (08.11.2017-71306642-050.01.04). The protocol conforms to CONSORT guidelines for parallel-group randomized trials and the protocol is designed to conform to the principles of the Declaration of Helsinki.

Participant :

The investigators will enroll 246 patients with primary bilateral symptomatic knee osteoarthritis that was refractory to conservative treatment who underwent bilateral TKA (total knee arthroplasty) under single anaesthesia between 2017 and 2018. An informed consent form will be obtained from all patients.

The schedule for randomization was randomly generated using a computer before the initiation of the trial. Patients were randomly assigned in a 1:1 ratio. A blind medical staff member will organize the days of the surgeries of randomized patients for the two-surgeon (TS) or single-surgeon (SS) groups. Neither patients nor assessors will know about randomization results. The outcome assessor will be blinded to group allocation and will no involve in providing the interventions. The statistician performing the statistical analyses will be blinded to group allocation.

Surgical procedures:

All surgeries will be performed by two high-volume surgeons under regional or general anaesthesia. Both surgeons always will operate on the same side. Each of patients will receive a total knee prostheses-Vanguard (Zimmer Biomet,Inc, Warsaw, IN) - using a standard medial parapatellar approach without the use of a tourniquet. All patients will be given 2 g cefazolin for infection prophylaxis and 1 g tranexamic acid for blood loss prophylaxis intravenously 30 min before the incision. In the TS group, the two surgeons will start the incisions at the same time using two different instrumentation sets and with their own scrub nurses. In the SS group, the surgeon will operate on both knees consecutively. No Hemovac drains will be used in either group. After closing the joint capsule, 1 g tranexamic acid will be injected into the joint in both groups.

All patients will start a standard physiotherapy program with the same blinded therapist. All patients will be started walking on the first postoperative day, using two crutches or a walker. Antibiotic prophylaxis will be continued for 24 h with 1 g intravenous cefazolin every 6 h. Venous thromboembolism prophylaxis will be administered using low-molecular-weight heparin for 4 weeks postoperatively. The investigators will check the estimated blood loss (EBL) on the first postoperative day. All patients will be asked to visit our outpatient clinic at 2 and 6 weeks and 3 months postoperatively. For functional outcomes and pain will be used the Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and a visual analog scale (VAS) preoperatively and 90 days postoperatively.

Primary Outcome:

The prespecified primary outcome was the between-group difference according to the rate of major complications.The investigators will assess major complications in all patients until 90 days postoperatively.

Secondary Outcomes:

The investigators also will assess the estimated blood loss (EBL), minor complications, operation time and functional results among the groups. The EBL will be calculated using the Gross formula and compared between the groups.

Statistical methods:

Categorical variables will be analyzed using the chi-square test and continuous variables will be tested using the Mann-Whitney U-test. The statistical analyses will be performed using IBM SPSS Statistics for Windows, ver. 22.0. (IBM, Armonk, NY). Significance was set at α < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Primary bilateral knee osteoarthritis with refractory to conservative treatment
* Patients who accept participation in the research and the randomization

Exclusion Criteria:

* no history of malignancy
* less than 75 years old
* without severe extra-articular deformities
* severe cardiac insufficiency and morbid obesity
* without systemic inflammatory diseases

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of major complications | 90 days
  Systemic and local major complications will evaluate. Major complications are conditions that require long-term hospitalization and repetitive intervention.

SECONDARY OUTCOMES:
Number of minor complications | 90 days
  Systemic and local minor complications will evaluate. Minor complications are conditions that require long-term hospitalization or requires strict follow-up.
WOMAC knee score | 90 days
  Score evaluating the patient's functional status before and after arthroplasty
Oxford Knee Score | 90 days
  Score evaluating the patient's functional status before and after arthroplasty
Estimated blood loss | 1 day after operation
  Estimated blood loss in post op 1 day by calculating with Gross formula

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uzer G, Aliyev O, Yildiz F, Gungoren N, Elmali N, Tuncay I. Safety of one-stage bilateral total knee arthroplasty -one surgeon sequential vs. two surgeons simultaneous: a randomized controlled study. Int Orthop. 2020 Oct;44(10):2009-2015. doi: 10.1007/s00264-020-04704-9. Epub 2020 Jul 10. PMID 32651711